CLINICAL TRIAL: NCT04118595
Title: Reducing the Transition From Acute to Chronic Musculoskeletal Pain Among Older Adults
Acronym: BETTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Duke University (Other); Indiana University (Other); Yale University (Other); Elon University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-0204; R01AG058702 (NIH)
Record Dates: First submitted 2019-09-27; First posted 2019-10-08 (Actual); Results first posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-08

CONDITIONS: Acute Musculoskeletal Pain; Chronic Pain
Keywords: Musculoskeletal Pain; Acute Pain; Emergency Department; Elderly; Video
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain; Acute Pain; Emergencies | interventions — Telemedicine; Physicians, Primary Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Full Intervention (Video + Telecare + PCP communication) (Experimental): Patients in this arm will watch an interactive pain management video; receive a pain assessment phone call and be given medication and behavioral pain management strategy recommendations; and an index visit and telecare summary will be shared with patient's primary care provider.
  Interventions: Behavioral: Educational Video; Behavioral: Telecare; Behavioral: Correspondence with Primary Care Provider
- Video-only Intervention (Experimental): Patients in this arm will watch an interactive pain management video.
  Interventions: Behavioral: Educational Video
- Usual Care (No Intervention): Patients will receive the typical care provided by medical personnel for their acute pain.

INTERVENTIONS:
Behavioral: Educational Video — Educational Video: Development of the original video was funded by the John A. Hartford Foundation and used a systematic approach that included a review of literature and current pain management guidelines and input from emergency physicians, geriatricians, and experts in pharmacology, physical therapy, and risk communication. The video offers information about the pharmacologic management of acute musculoskeletal pain (MSP) and recovery-promoting behaviors. Each video section is followed by a multiple-choice question to promote interaction and reinforce learning. The actress for the 13-minute video is a 56-year-old mixed-race woman who presents herself as a healthcare provider. The video script was developed for a grade level 5.5 and will be shown to the patient within 24 hours of the acute care visit. A link to the video is emailed or texted to the patient.
  Arms: Full Intervention (Video + Telecare + PCP communication); Video-only Intervention
Behavioral: Telecare — Telecare will be provided via a protocol-guided phone call from a nurse care manager 48-72 hours after discharge from the ED or orthopedic urgent care. The call is designed to support patient decision-making regarding analgesics and behaviors following the content presented in the video. Topics covered in the call will include discussion of goals and priorities the patient has for their pain management, current prescriptions and analgesic use (and adjustments if needed), non-pharmacologic methods of pain management, warnings about potential side effects, current healthcare utilization, and open-ended questions to address additional patient care needs. Conversations will be guided by a shared decision making framework in which the nurse suggests pain management options, discusses their pros and cons, and actively elicits feedback from the patient. The telecare call is designed to last 15 minutes.
  Arms: Full Intervention (Video + Telecare + PCP communication)
Behavioral: Correspondence with Primary Care Provider — Following the telecare conversation, a note will be sent directly to the patient's primary care provider using a secure email or an electronic message that includes: 1) The date, time, location and reason for the index visit; (2) Results of diagnostics studies; (3) Discharge prescriptions/ recommendations; (4) A summary of and link to the video, explaining the emphasis on patient knowledge and SDM; (5) A summary of the telecare conversation; and (6) Encouragement for follow-up. PCPs will be asked to confirm receipt of this message.
  Arms: Full Intervention (Video + Telecare + PCP communication)

SUMMARY:
The investigators have developed a three component intervention to support shared decision-making during the early recovery phase for older adults who present to the emergency department (ED) or orthopedic urgent care with acute musculoskeletal pain. The first component is a brief interactive video to enhance patient knowledge and self-efficacy regarding treatment options with the intent of facilitating conversations between patients and emergency providers. The second component is a protocol-guided phone conversation (telecare) between a nurse care manager and the patient at 48-72 hours following discharge to assess pain severity and interference with daily activities, review analgesic use and side effects and recovery-promoting behaviors, and discuss adjustments to the patients treatment. The third component is communication with the patient's primary care provider following the telecare call to inform them of the patient's condition and treatment plan and encourage primary care followup. The short-term objective of this project is to test the efficacy of this intervention to reduce the transition from acute to chronic musculoskeletal pain among older adults and obtain data to inform implementation. The investigators will conduct a three-arm randomized controlled trial with adults aged 50 years and older who present to the ED or orthopedic urgent care with acute musculoskeletal pain. Patients will be randomized to (1) the full intervention (video + telecare + communication with primary provider), (2) video alone, or (3) usual care. The primary outcome will be pain, measured longitudinally over the course of the year following the acute care visit. Secondary outcomes will include physical function, analgesic side effects and adverse events, opioid use, depression and anxiety symptoms, sleep duration and quality, and healthcare utilization at one, three, six, and twelve months. Secondary analyses will (1) examine whether the intervention has its effect by promoting shared decision-making, and (2) estimate the cost-effectiveness of the intervention. The long-term goal of this work is to develop, test, and implement interventions that improve long-term health outcomes for older adults with acute musculoskeletal pain.

DETAILED DESCRIPTION:
Participants will be assigned to one of the three treatment arms using 1:1:1 randomization, stratified by access to a primary care provider, using randomly permuted blocks with random block sizes. (Primary care access will be determined using Source of Care questions from the Primary Care Assessment tool.) Randomization will be based on computer generated lists and allocated within subgroups based on access to a PCP using REDCap's integrated randomization module. One arm will receive the full intervention (educational video, telecare call, transmission of clinical information to the PCP), one will view the educational video only, and one will receive usual care. The investigators decided against a 2x2 factorial design, which would add a telecare only arm, because our team' s collective understanding is that a basic understanding of pain management (as provided by the educational video) is essential for effective shared decision-making (SDM) and often missing among older patients. Screening, consent, randomization, and assessments will be completed by the study coordinator.

Interventions

Educational Video: Development of the original video was funded by the John A. Hartford Foundation and used a systematic approach that included a review of literature and current pain management guidelines and input from emergency physicians, geriatricians, and experts in pharmacology, physical therapy, and risk communication. The video offers information about the pharmacologic management of acute musculoskeletal pain (MSP) and recovery-promoting behaviors. Each video section is followed by a multiple-choice question to promote interaction and reinforce learning. The actress for the 13-minute video is a 56-year-old mixed-race woman who presents herself as a healthcare provider. The video script was developed for a grade level 5.5 and will be shown to the patient within 24 hours of the acute care visit. A link to the video is emailed or texted to the patient.

Telecare: Telecare will be provided via a protocol-guided phone call from a nurse care manager 48-72 hours after discharge. The call is designed to support patient decision-making regarding analgesics and behaviors following the content presented in the video. Before the call, the nurse will review the note from the index visit to obtain information about comorbidities, medications, allergies, and the patient's evaluation and treatment in the ED. Topics covered in the call will include discussion of pain management goals and priorities, current analgesic use, non-pharmacologic methods of pain management, warnings about potential side effects, and open-ended questions to address additional patient care needs. Conversations will be guided by an SDM framework in which the nurse elicits information from the patient, then discusses with the patient alternative strategies, and actively elicits feedback from the patient. Patients will be encouraged to follow-up with their PCP; uninsured patients will be referred to local free or low-cost medical clinics. The telecare call is designed to last 15 minutes and the nurse will be trained to complete the call in 15 minutes.

Correspondence with PCP: Following the telecare conversation, the nurse will enter a note in the Electronic Health Record (EHR) documenting the patient's current clinical status, information reviewed, and any recommendations or referrals made. The nurse will then share this note directly with the patient's PCP using a secure e-mail or an electronic message within the EHR if the PCP is a University of North Carolina (UNC)-affiliated provider. (If the PCP's email address is not available, the research staff will contact the PCP or their office by phone to obtain an email address or fax number.) This communication with also include: (1) The date, time, location and reason for the initial visit; (2) Results of diagnostics studies; (3) Discharge prescriptions/recommendations; (4) A summary of and link to the video, explaining the emphasis on patient knowledge and SDM; (5) summary of the telecare conversation; and (6) encouragement for follow-up. PCPs will be asked to confirm receipt of this message.

*Study outcome measures as described in this CT.gov report have been revised as of September 6, 2023 in order to reflect the final Master Protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years and older
* Present to UNC ED patient with primary complaint of acute musculoskeletal pain
* Average pain score >/= 4 on 0-10 scale
* Expected discharge from the ED

Exclusion Criteria:

* patient does not speak English
* primary pain located in the head, chest, or abdomen
* pain due to ischemia, infection, or some other cause not due to MSP (blood clot, kidney stone, etc.)
* primary pain due to self-injury
* patient is critically ill determined by an acuity score of 1 in the tracking board
* diagnosis of somatoform disorder, schizophrenia, dementia, or bipolar disorder
* patient is a prisoner or in police custody
* self-reported daily opioid use for more than 2 weeks
* resides in a nursing home or is homeless
* at-risk alcohol use
* speech, hearing, vision problems
* cognitively impaired (6-item Brief Screener)
* nonworking phone number (follow-up occurs via phone calls)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2023-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Meyer, PhD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Hospitals, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with The University of North Carolina.
Time Frame: Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication.
Access Criteria: Investigator who proposes data use has approval from an IRB, IEC, or REB, as applicable, and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Background] Platts-Mills TF, Hollowell AG, Burke GF, Zimmerman S, Dayaa JA, Quigley BR, Bush M, Weinberger M, Weaver MA. Randomized controlled pilot study of an educational video plus telecare for the early outpatient management of musculoskeletal pain among older emergency department patients. Trials. 2018 Jan 5;19(1):10. doi: 10.1186/s13063-017-2403-8. PMID 29304831
- [Background] Gan TJ, Joshi GP, Zhao SZ, Hanna DB, Cheung RY, Chen C. Presurgical intravenous parecoxib sodium and follow-up oral valdecoxib for pain management after laparoscopic cholecystectomy surgery reduces opioid requirements and opioid-related adverse effects. Acta Anaesthesiol Scand. 2004 Oct;48(9):1194-207. doi: 10.1111/j.1399-6576.2004.00495.x. PMID 15352969
- [Background] Hurka-Richardson K, Platts-Mills TF, McLean SA, Weinberger M, Stearns SC, Bush M, Quackenbush E, Chari S, Aylward A, Kroenke K, Kerns RD, Weaver MA, Keefe FJ, Berkoff D, Meyer ML. Brief Educational Video plus Telecare to Enhance Recovery for Older Emergency Department Patients with Acute Musculoskeletal Pain: an update to the study protocol for a randomized controlled trial. Trials. 2022 May 12;23(1):400. doi: 10.1186/s13063-022-06310-z. PMID 35550175
- [Derived] Platts-Mills TF, McLean SA, Weinberger M, Stearns SC, Bush M, Teresi BB, Hurka-Richardson K, Kroenke K, Kerns RD, Weaver MA, Keefe FJ. Brief educational video plus telecare to enhance recovery for older emergency department patients with acute musculoskeletal pain: study protocol for the BETTER randomized controlled trial. Trials. 2020 Jul 6;21(1):615. doi: 10.1186/s13063-020-04552-3. PMID 32631400

RESULTS

PARTICIPANT FLOW:
Groups:
- Full Intervention (Video + Telecare + PCP Communication): Patients in this arm will watch an interactive pain management video; receive a pain assessment phone call and be given medication and behavioral pain management strategy recommendations; and an index visit and telecare summary will be shared with patient's primary care provider.
  Educational Video: The video offers information about the pharmacologic management of acute musculoskeletal pain (MSP) and recovery-promoting behaviors. Each video section is followed by a multiple-choice question to promote interaction and reinforce learning. The video script was developed for a grade level 5.5 and will be shown to the patient within 24 hours of the acute care visit. A video link is emailed or texted to the patient.
  Telecare: Telecare will be provided via a protocol-guided phone call from a nurse care manager 48-72 hours after discharge from the emergency department (ED) or orthopedic urgent care. The call is designed to support patient decision-making regarding analgesics and behaviors following the content presented in the video.
  Correspondence with Primary Care Provider: Following the telecare conversation, a note will be sent directly to the patient's primary care provider using a secure email that includes: 1) The date, time, location and reason for the index visit; (2) Results of diagnostics studies; (3) Discharge prescriptions/ recommendations; (4) A summary of and link to the video; (5) A summary of the telecare conversation; and (6) Encouragement for follow-up.
- Video-only Intervention: Patients in this arm will watch an interactive pain management video.
  Educational Video: The video offers information about the pharmacologic management of acute musculoskeletal pain (MSP) and recovery-promoting behaviors. Each video section is followed by a multiple-choice question to promote interaction and reinforce learning. The video script was developed for a grade level 5.5 and will be shown to the patient within 24 hours of the acute care visit. A link to the video is emailed or texted to the patient.
Period: Overall Study
Arm/Group | Full Intervention (Video + Telecare + PCP Communication) | Video-only Intervention | Usual Care
Started | 112 | 107 | 111
Completed Week 1 Within 7-day Window | 107 | 97 | 108
Completed Month 1 Within 7-day Window | 108 | 100 | 106
Completed Month 3 Within 7-day Window | 103 | 99 | 102
Completed Month 6 Within 7-day Window | 104 | 96 | 102
Completed Month 12 Within 7-day Window | 101 | 88 | 96
Completed | 101 | 88 | 96
Not Completed | 11 | 19 | 15

BASELINE CHARACTERISTICS:
Groups:
- Full Intervention (Video + Telecare + PCP Communication): Patients in this arm will watch an interactive pain management video; receive a pain assessment phone call and be given medication and behavioral pain management strategy recommendations; and an index visit and telecare summary will be shared with patient's primary care provider.
  Educational Video: The video offers information about the pharmacologic management of acute musculoskeletal pain (MSP) and recovery-promoting behaviors. Each video section is followed by a multiple-choice question to promote interaction and reinforce learning. The video script was developed for a grade level 5.5 and will be shown to the patient within 24 hours of the acute care visit. A link to the video is emailed or texted to the patient.
  Telecare: Telecare will be provided via a protocol-guided phone call from a nurse care manager 48-72 hours after discharge from the ED or orthopedic urgent care. The call is designed to support patient decision-making regarding analgesics and behaviors following the content presented in the video.
  Correspondence with Primary Care Provider: Following the telecare conversation, a note will be sent directly to the patient's primary care provider using a secure email that includes: 1) The date, time, location and reason for the index visit; (2) Results of diagnostics studies; (3) Discharge prescriptions/ recommendations; (4) A summary of and link to the video; (5) A summary of the telecare conversation; and (6) Encouragement for follow-up.
- Total: Total of all reporting groups
Arm/Group | Full Intervention (Video + Telecare + PCP Communication) | Video-only Intervention | Usual Care | Total
Number analyzed (Participants) | 112 | 107 | 111 | 330
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (9.9) | 65.1 (8.8) | 64.4 (8.7) | 64.7 (9.1)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years old | 60 | 58 | 59 | 177
  65 years old or greater | 52 | 49 | 52 | 153
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 72 | 72 | 226
  Male | 30 | 35 | 39 | 104
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 4 | 11
  Not Hispanic or Latino | 108 | 104 | 107 | 319
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 17 | 17 | 18 | 52
  White | 83 | 74 | 82 | 239
  More than one race | 0 | 1 | 2 | 3
  Unknown or Not Reported | 9 | 14 | 9 | 32
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 112 | 107 | 111 | 330

OUTCOME MEASURES:

1. Primary Outcome: Mean Brief Pain Inventory-Short Form (BPI-SF) Combined Pain Severity and Interference Score
Description: The Brief Pain Inventory-Short Form (BPI-SF) is an 11-item measure of pain severity and pain interference. Patients will rate their pain severity and interference over the past week on a 0-10 numeric scale at 3 discrete time periods (1, 3, and 6 months). End points for the severity items include 0 which equals "no pain" and 10 which equals "pain as bad as you can imagine." End points for the interference items include 0 which equals "does not interfere" and 10 "completely interferes." Higher scores reflect more pain severity and more pain interference. A composite score will be calculated by averaging scores from both the pain severity and interference items (all 11-items). Results from the 3 time periods will be analyzed longitudinally.
Time Frame: Month 1 (following ED or orthopedic urgent care visit) to Month 6
Population: Data are reported for all participants who completed each Follow-up within the 7-day window. There was participant attrition over time as shown in the Participant Flow.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Full Intervention (Video + Telecare + PCP Communication) | Video-only Intervention | Usual Care
Number analyzed (Participants) | 108 | 100 | 106
score on a scale
  Month 1 | 2.67 (2.09) | 2.99 (2.12) | 2.94 (2.29)
  Month 3: number analyzed (Participants) | 103 | 99 | 102
  Month 3 | 1.90 (1.80) | 2.18 (2.15) | 2.57 (2.34)
  Month 6: number analyzed (Participants) | 104 | 96 | 102
  Month 6 | 2.22 (2.21) | 2.35 (2.46) | 2.84 (2.41)
Statistical Analysis 1: Comparison: Full Intervention (Video + Telecare + PCP Communication) vs Video-only Intervention vs Usual Care; Test type: Superiority; p = 0.13, ANCOVA

2. Secondary Outcome: Mean Pain Severity on the Brief Pain Inventory-Short Form (BPI-SF) Score
Description: The BPI-SF is an 11-item measure of pain severity and pain interference with severity entailing 4 of the questions. Patient's will rate their pain severity over the past week on a 0-10 numeric rating scale, with a higher score reflecting more pain. End points include 0 which equals "no pain" and 10 which equals "pain as bad as you can imagine." Answers to each of the 4 questions will be reported as mean values for each time point (Month 1, 3, and 6).
Time Frame: Up to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Full Intervention (Video + Telecare + PCP Communication) | Video-only Intervention | Usual Care
Number analyzed (Participants) | 108 | 100 | 106
score on a scale
  Month 1 | 2.69 (2.00) | 2.94 (1.97) | 2.90 (2.14)
  Month 3: number analyzed (Participants) | 103 | 99 | 102
  Month 3 | 1.98 (1.79) | 2.22 (2.10) | 2.53 (2.25)
  Month 6: number analyzed (Participants) | 104 | 96 | 102
  Month 6 | 2.30 (2.14) | 2.45 (2.42) | 2.81 (2.27)
Statistical Analysis 1: Comparison: Full Intervention (Video + Telecare + PCP Communication) vs Video-only Intervention vs Usual Care; Test type: Superiority; p = 0.41, ANCOVA

3. Secondary Outcome: Mean Pain Interference on the BPI-SF Score
Description: The BPI-SF is an 11-item measure of pain severity and pain interference with interference with daily activities entailing 7 of the questions. Patient's will rate their pain interference over the past week, on a 0-10 scale with a higher score reflecting more interference with activities. End points include 0 which equals "does not interfere" and 10 which equals "completely interferes." Answers to each of the 7 questions will be reported as mean values for each time point (Month 1, 3, and 6).
Time Frame: Up to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Full Intervention (Video + Telecare + PCP Communication) | Video-only Intervention | Usual Care
Number analyzed (Participants) | 108 | 100 | 106
score on a scale
  Month 1 | 2.64 (2.40) | 3.04 (2.51) | 2.98 (2.70)
  Month 3: number analyzed (Participants) | 103 | 99 | 102
  Month 3 | 1.82 (1.99) | 2.14 (2.38) | 2.61 (2.64)
  Month 6: number analyzed (Participants) | 104 | 96 | 102
  Month 6 | 2.14 (2.43) | 2.26 (2.72) | 2.88 (2.76)
Statistical Analysis 1: Comparison: Full Intervention (Video + Telecare + PCP Communication) vs Video-only Intervention vs Usual Care; Test type: Superiority; p = 0.08, ANCOVA

4. Secondary Outcome: Mean Symptom Distress Score
Description: The Opioid-Related Symptom Distress Scale (OR-SDS) will be used to assess subject-reported levels of frequency and severity of 10 symptoms known to be associated with opioid medication usage, such as drowsiness, dizziness, and constipation. Added to this measure are 5 other symptoms (including shortness of breath, falls, abdominal pain, bloody stool, and 'other'), reflecting side effects for patients taking NSAIDs or acetaminophen. Symptom frequency will be rated as: 1=rarely, 2=occasionally, 3=frequently, or 4=almost constantly, with higher ratings indicating more frequent symptoms (ranging from 1 to 4). Symptom severity will be rated as: 1=slightly, 2-moderate, 3=severe, or 4=very severe, with higher ratings indicating more severe symptoms (ranging from 1 to 4). Patients who deny a symptom will be given a score of zero for frequency and severity. A mean symptom distress score was calculated for each arm based on patient reported scores for severity and frequency.
Time Frame: 1 week & 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Full Intervention (Video + Telecare + PCP Communication) | Video-only Intervention | Usual Care
Number analyzed (Participants) | 108 | 100 | 108
score on a scale
  Week 1: number analyzed (Participants) | 107 | 97 | 108
  Week 1 | 0.062 (0.138) | 0.063 (0.164) | 0.043 (0.103)
  Month 1: number analyzed (Participants) | 108 | 100 | 106
  Month 1 | 0.023 (0.080) | 0.019 (0.065) | 0.015 (0.058)
Statistical Analysis 1: Comparison: Full Intervention (Video + Telecare + PCP Communication) vs Video-only Intervention vs Usual Care; Test type: Superiority; p = 0.64, ANCOVA

5. Secondary Outcome: Percent of Participants With Opioid Use During the Past Week
Description: Patients will be asked if they have used opioids during the past week at each of the follow-up time points. This will be a dichotomous outcome in which 'yes' will indicate opioid use in the past week and 'no' will indicate no opioid use in the past week.
Time Frame: 1, 3, 6, and 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Full Intervention (Video + Telecare + PCP Communication) | Video-only Intervention | Usual Care
Number analyzed (Participants) | 108 | 100 | 106
percentage of participants
  Month 1-Yes | 5.6 | 9.0 | 5.7
  Month 3-Yes: number analyzed (Participants) | 103 | 99 | 102
  Month 3-Yes | 1.9 | 1.0 | 4.9
  Month 6-Yes: number analyzed (Participants) | 104 | 96 | 102
  Month 6-Yes | 2.9 | 3.1 | 5.9
  Month 12-Yes: number analyzed (Participants) | 100 | 88 | 96
  Month 12-Yes | 3.0 | 3.4 | 6.3
Statistical Analysis 1: Comparison: Full Intervention (Video + Telecare + PCP Communication) vs Video-only Intervention vs Usual Care; Test type: Superiority; p = 0.57, ANCOVA

6. Secondary Outcome: PROMIS Measure: Mean T-score Physical Function-4
Description: Patient report of physical function will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function-4 for chores, ability to use stairs, walking, and running errands on a 5-point scale with end points of "without any difficulty" and "unable to do." Higher scores reflect less difficulty. T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points. Therefore a person with a T-score of 40 is one SD below the mean. These values will be compared to the value obtained from the baseline assessment with patients reporting their function prior to injury. The data will be analyzed longitudinally for months 1, 3, 6, and 12 (following the approach for BPI for the primary outcome).
Time Frame: 1, 3, 6, and 12 months
Population: Data are reported for all participants who completed each Follow-up within the 7-day window. There was participant attrition over time as shown in the Participant Flow. One participant in the Full Intervention (Video + Telecare + PCP communication) arm did not complete the 3 month assessment.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Full Intervention (Video + Telecare + PCP Communication) | Video-only Intervention | Usual Care
Number analyzed (Participants) | 108 | 100 | 106
T-score
  Month 1 | 42.19 (8.10) | 40.83 (8.26) | 41.17 (8.54)
  Month 3: number analyzed (Participants) | 102 | 99 | 102
  Month 3 | 45.25 (8.23) | 44.21 (8.51) | 43.49 (9.26)
  Month 6: number analyzed (Participants) | 104 | 96 | 102
  Month 6 | 45.88 (9.00) | 44.41 (8.98) | 43.51 (9.23)
  Month 12: number analyzed (Participants) | 101 | 88 | 96
  Month 12 | 47.44 (8.54) | 46.29 (8.94) | 44.50 (9.54)
Statistical Analysis 1: Comparison: Full Intervention (Video + Telecare + PCP Communication) vs Video-only Intervention vs Usual Care; Test type: Superiority; p = 0.43, ANCOVA

7. Secondary Outcome: PROMIS Measure: Mean T-score Global Health-Physical 2a
Description: Patient reported global health will be measured using the PROMIS Global Health-Physical 2a. General physical health is measured on a 5-point scale with end points of "excellent" and "poor," where higher scores reflect better physical health. Ability to carry out every day physical activities is measured on a 5 point scale with end points of "completely" and "not at all," where higher scores reflect better ability. T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points. Therefore a person with a T-score of 40 is one SD below the mean. These values will be compared to the value obtained from the baseline assessment with patients reporting their global health prior to injury. The data will be analyzed longitudinally for months 1, 3, 6, and 12 (following the approach for BPI for the primary outcome).
Time Frame: 1, 3, 6, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Full Intervention (Video + Telecare + PCP Communication) | Video-only Intervention | Usual Care
Number analyzed (Participants) | 108 | 100 | 106
T-score
  Month 1 | 47.73 (7.89) | 45.72 (7.54) | 46.75 (8.24)
  Month 3: number analyzed (Participants) | 103 | 99 | 102
  Month 3 | 49.67 (7.14) | 48.55 (8.14) | 47.47 (9.42)
  Month 6: number analyzed (Participants) | 104 | 96 | 102
  Month 6 | 49.68 (8.91) | 47.87 (8.69) | 47.52 (8.89)
  Month 12: number analyzed (Participants) | 101 | 88 | 96
  Month 12 | 50.08 (7.92) | 49.16 (8.69) | 47.78 (8.58)
Statistical Analysis 1: Comparison: Full Intervention (Video + Telecare + PCP Communication) vs Video-only Intervention vs Usual Care; Test type: Superiority; p = 0.19, ANCOVA

8. Secondary Outcome: Healthcare Utilization, Mean Days in the Hospital
Description: The number of days the patient spent in the hospital after ED discharge will be collected through patient report and the patient's electronic health record. Analysis will compare these outcomes among study arms.
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Full Intervention (Video + Telecare + PCP Communication) | Video-only Intervention | Usual Care
Number analyzed (Participants) | 108 | 100 | 106
Days
  Month 1 | 0.04 (0.30) | 0.00 (0.00) | 0.05 (0.29)
  Month 3: number analyzed (Participants) | 103 | 99 | 102
  Month 3 | 0.16 (1.22) | 0.01 (0.10) | 0.10 (0.67)
  Month 6: number analyzed (Participants) | 104 | 96 | 102
  Month 6 | 0.00 (0.00) | 0.07 (0.62) | 0.17 (1.23)
  Month 12: number analyzed (Participants) | 101 | 88 | 96
  Month 12 | 0.23 (1.09) | 0.09 (0.39) | 0.13 (0.39)
Statistical Analysis 1: Comparison: Full Intervention (Video + Telecare + PCP Communication) vs Video-only Intervention vs Usual Care; Test type: Superiority; p = 0.15, ANCOVA

9. Secondary Outcome: Healthcare Utilization, Mean Number of Visits to ED/Urgent Care
Description: The number of visits to an ED or urgent care will be collected through patient report and the patient's electronic health record. Analysis will compare these outcomes among study arms.
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Full Intervention (Video + Telecare + PCP Communication) | Video-only Intervention | Usual Care
Number analyzed (Participants) | 108 | 100 | 106
visits
  Month 1 | 0.09 (0.35) | 0.06 (0.24) | 0.04 (0.19)
  Month 3: number analyzed (Participants) | 103 | 99 | 102
  Month 3 | 0.25 (0.85) | 0.08 (0.31) | 0.25 (0.62)
  Month 6: number analyzed (Participants) | 104 | 96 | 102
  Month 6 | 0.30 (1.45) | 0.26 (0.71) | 0.40 (1.08)
  Month 12: number analyzed (Participants) | 101 | 88 | 96
  Month 12 | 0.40 (1.21) | 0.35 (0.76) | 0.35 (0.74)
Statistical Analysis 1: Comparison: Full Intervention (Video + Telecare + PCP Communication) vs Video-only Intervention vs Usual Care; Test type: Superiority; p = 0.04, ANCOVA

10. Secondary Outcome: Healthcare Utilization, Mean Number of Visits to Primary Care Provider
Description: The number of visits to a primary care provider's office will be collected through patient report and the patient's electronic health record. Analysis will compare these outcomes among study arms.
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Full Intervention (Video + Telecare + PCP Communication) | Video-only Intervention | Usual Care
Number analyzed (Participants) | 108 | 100 | 106
visits
  Month 1 | 0.15 (0.43) | 0.22 (0.48) | 0.17 (0.42)
  Month 3: number analyzed (Participants) | 103 | 99 | 102
  Month 3 | 0.50 (0.78) | 0.42 (0.86) | 0.53 (0.77)
  Month 6: number analyzed (Participants) | 104 | 96 | 102
  Month 6 | 0.70 (0.82) | 0.79 (1.05) | 0.81 (0.96)
  Month 12: number analyzed (Participants) | 101 | 88 | 96
  Month 12 | 1.50 (1.73) | 1.10 (1.12) | 1.39 (1.35)
Statistical Analysis 1: Comparison: Full Intervention (Video + Telecare + PCP Communication) vs Video-only Intervention vs Usual Care; Test type: Superiority; p = 0.36, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent to study exit, up to 12 months.
Arm/Group | Full Intervention (Video + Telecare + PCP Communication) | Video-only Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/112 | 1/107 | 1/111
Serious Adverse Events (participants affected / at risk) | 6/112 | 3/107 | 13/111
Other Adverse Events (participants affected / at risk) | 38/112 | 39/107 | 35/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Full Intervention (Video + Telecare + PCP Communication) (N=112) | Video-only Intervention (N=107) | Usual Care (N=111)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2)
Bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Endocarditis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Leukemia secondary to oncology chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) — Based on study suicide assessment
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Full Intervention (Video + Telecare + PCP Communication) (N=112) | Video-only Intervention (N=107) | Usual Care (N=111)
Abdominal pain (Gastrointestinal disorders) | 4 (7) | 7 (9) | 7 (7)
Constipation (Gastrointestinal disorders) | 5 (9) | 7 (7) | 11 (13)
Fatigue (General disorders) | 12 (14) | 10 (11) | 8 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2) | 8 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (15) | 10 (10) | 6 (8)
Concentration impairment (Nervous system disorders) | 7 (8) | 3 (3) | 3 (3)
Dizziness (Nervous system disorders) | 6 (6) | 2 (2) | 3 (3)
Somnolence (Nervous system disorders) | 17 (20) | 16 (17) | 14 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2023-09-12): https://cdn.clinicaltrials.gov/large-docs/95/NCT04118595/Prot_002.pdf
  • Statistical Analysis Plan (2022-07-24): https://cdn.clinicaltrials.gov/large-docs/95/NCT04118595/SAP_003.pdf
  • Informed Consent Form (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/95/NCT04118595/ICF_001.pdf